CLINICAL TRIAL: NCT04803175
Title: Prospective Comparison of Sacubitril/Valsartan Versus Valsartan on the Outcome of Heart Failure With Improved Ejection Fraction: a Pilot Study
Brief Title: Sacubitril/Valsartan Versus Valsartan in Heart Failure With Improved Ejection Fraction
Acronym: PROSPER-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Oh Choi, Division of Cardiology, Department of Medicine, Heart Vascular Stroke Institute, Samsung Medical Center
Other Study IDs: 2020-08-082
Record Dates: First submitted 2021-02-25; First posted 2021-03-17 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure, Systolic
Keywords: Heart Failure with reduced Ejection Fraction; Heart Failure with improved Ejection Fraction; Sacubitril/valsartan; Valsartan
MeSH Terms: conditions — Heart Failure, Systolic | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sacubitril/valsartan: Patients undergoing continued treatment with sacubitril/valsartan after improvement of LVEF >40% with > 3 months of sacubitril/valsartan treatment. Dose and titration schedule will be individualized by discretion of the attending physician.
  Interventions: Drug: Sacubitril-Valsartan
- Valsartan: Patients undergoing continued treatment with valsartan after improvement of LVEF >40% with > 3 months of sacubitril/valsartan treatment. Dose and titration schedule will be individualized by discretion of the attending physician.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Participants will receive individualized dosage and titration as part of routine medical care, and a the effect will be studied for at least 12 months. The investigator does not assign specific interventions to the study participants.
  Other Names: Entresto
  Groups: Sacubitril/valsartan
Drug: Valsartan — Participants will receive individualized dosage and titration as part of routine medical care, and a the effect will be studied for at least 12 months. The investigator does not assign specific interventions to the study participants.
  Other Names: Diovan
  Groups: Valsartan

SUMMARY:
Heart failure (HF) is a chronic disease with weakened heart muscles or abnormal pressure within the heart chambers result in breathlessness, leg edema, or fatigue. A subclass of HF shows reduced heart muscle contractility, which is represented by the left ventricular ejection fraction (LVEF). Valsartan is an angiotensin II receptor blocker, a major drug class for heart failure. Sacubitril/valsartan is a combination of 2 drugs, classified as a new class of drug called angiotensin receptor neprilysin inhibitor (ARNI). Although these medications are both first-line treatment in HF with reduced LVEF, recent guidelines encourage the use of sacubitril/valsartan in patients with ongoing symptoms. After successful treatment, some patients experience recovery of LVEF. In these patients, otherwise called heart failure with improved ejection fraction (HFiEF), it is not clear whether continued treatment with sacubitril/valsartan or valsartan is beneficial in terms of relapse of heart failure or worsening of LVEF. Therefore, the investigators aim to determine whether the treatment with sacubitril/valsartan versus valsartan differs in clinical outcomes after 1 year in HFiEF patients by observing the change in blood test markers of heart failure (N-terminal prohormone of brain natriuretic peptide; NT-proBNP) and aggravation of HF defined as reduced LVEF, congestive symptoms, hospitalization or death from HF.

DETAILED DESCRIPTION:
1. Background and study purpose Heart failure (HF) is caused by structural or functional abnormality of the myocardium or elevated intracardiac pressures, resulting in symptoms and signs of low cardiac output or congestion, such as dyspnea, peripheral edema, elevated jugular venous pressures, pulmonary congestion, and fatigue. HF with reduced left ventricular ejection fraction (HFrEF) is defined as an LVEF <40% by the 2013 American College of Cardiology/American Heart Association (ACC/AHA) guidelines. Recent guidelines recommend the use of angiotensin-converting enzyme inhibitors (ACEI)/angiotensin II receptor blocker (ARB)/angiotensin receptor neprilysin inhibitor (ARNI), beta blockers (BB), aldosterone antagonists (AA), and sodium-glucose co-transporter-2 inhibitors (SGLT2i) in HFrEF patients. ACEI/ARB/ARNI, collectively known as renin-angiotensin-system (RAS) blockers, are considered the most important drug class in the treatment for HFrEF and recently, ARNI is increasingly preferred as the first-choice drug. Unlike for initial treatment of HFrEF, continued treatment for patients who experience recovery of LVEF is not as well established. In these patients, called heart failure with improved ejection fraction (HFiEF), it is not clear whether continued treatment with sacubitril/valsartan or valsartan is beneficial in terms of relapse of heart failure or worsening of LVEF. Therefore, the investigators aim to determine whether the treatment with sacubitril/valsartan versus valsartan differs in clinical outcomes after 1 year in HFiEF patients by observing the change in serum N-terminal prohormone of brain natriuretic peptide (NT-proBNP) and clinical relapse of HF.

2. Registry factors

1. Source data verification will be done by comparing the data to electronic medical records and paper and electronic case report forms.
2. Data dictionary with detailed description of each variables are given.
3. Sample size assessment was calculated by comparing mean NT-proBNP levels at baseline and after 12 months in the two groups by two-sample t-test (two-sided, effect size=0.6, type I error=0.05, type II error=0.8, allocation ratio=1). With a drop-out rate of 10%, 50 patients in each group are needed. As the change of NT-proBNP in HFiEF with sacubitril/valsartan or valsartan has rarely been reported, estimation from the TRED-HF study (Lancet. 2019 Jan 5; 393(10166):61) was used as reference for effect size. This reference was a small study of 25 patients in each group. Therefore, the effect size used for calculation was modified to 0.6 rather than 0.8 by intuition of the investigators.
4. Plan for missing data: To avoid unavailable data, clinical visits will be monitored and calls will be made for missed appointments. Uninterpretable or out-of-range results will be discussed by participating investigators through regular meetings.
5. Statistical analysis Based on intention-to-treat analysis, the primary outcome (NT-proBNP changes) will be log-transformed and compared by paired t-tests. Baseline characteristics will be presented according to initial drug assignment and compared with the Mann-Whitney test for continuous variables or Fisher's exact test for categorical variables. Data are presented as median and IQR or as n (%). Occurrence of the secondary endpoint will be graphically displayed per group with Kaplan-Meier survival plots and compared with the log-rank test. Cox proportional hazards models will be used to investigate predictors of worsening NT-proBNP levels or occurrence of clinical adverse events in patients of each group. A p value less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria: (AND)

* Patient with a history of HF with reduced EF (HFrEF; LVEF <40 percent) and received treatment with sacubitril/valsartan for at least 3 months, after which showing improvement of LVEF to >40 percent and symptoms of NYHA functional class I or II
* serum NT-proBNP levels < 400 pg/dL for sinus rhythm and < 600pg/dL for atrial fibrillation
* Patients on stable doses of diuretics for 1 week

Exclusion Criteria: (OR)

* History of hospitalization for heart failure within 30 days before enrollment
* History of acute coronary syndrome (acute myocardial infarction or unstable angina), percutaneous coronary artery intervention or cardiac surgery within 30 days before enrollment
* History of cardiac resynchronization therapy within 90 days before screening
* Planned percutaneous or surgical coronary artery revascularization, or major cardiac surgery (coronary artery bypass, valvuloplasty, mechanical cardiac support or heart transplantation) within 90 days after enrollment
* Contraindicated or has history of hypersensitivity to RAS blockers including ACEI or ARB
* Use of inotropes
* Survival estimate < 3months
* Otherwise deemed as inappropriate by the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Consecutive participant sampling was done for all eligible patients.
  2. Patients visiting a specialized heart failure clinic at one of the top tertiary level hospitals in Seoul, Korea. Patients have a nationwide distribution geographically, and show a wide range of clinical presentations.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP concentration | Baseline, 6 months, 12 months
  pg/ml

SECONDARY OUTCOMES:
Heart failure relapse | 6 months and 12 months
  One or more of the following:
  1. LVEF <40 percent by cardiac imaging including but not refined to: echocardiography, cardiac magnetic resonance imaging
  2. symptomatic congestive heart failure: symptoms and signs of heart failure such as dyspnea, edema, abdominal fullness, and fatigue
Hospitalization for heart failure (HHF) | 6 months and 12 months
  Hospitalization for acute decompensated heart failure
Death caused by heart failure | 6 months and 12 months
  Heart failure being either the immediate or contributing cause of death.
Mortality | 6 months and 12 months
  All-cause mortality

OTHER OUTCOMES:
left ventricular (LV) ejection fraction (LVEF, percent) | 6 months (optional, personalized) and 12 months
  measurement based on echocardiography with the following priority
  1. Modified Simpson's method
  2. Visual estimation by a qualified echocardiography specialist
  3. M-mode
LV end-systolic dimension (LVESD, mm) | 6 months (optional, personalized) and 12 months
  measurement based on echocardiography with the following priority
  1. M-mode from parasternal long-axis view
  2. 2-d caliper from parasternal long-axis view
  3. M-mode from parasternal short-axis view
  4. 2-d caliper from parasternal short-axis view
  5. 2-d caliper from any other view
LV end-diastolic dimension (LVEDD, mm) | 6 months (optional, personalized) and 12 months
  measurement based on echocardiography with the following priority
  1. M-mode from parasternal long-axis view
  2. 2-d caliper from parasternal long-axis view
  3. M-mode from parasternal short-axis view
  4. 2-d caliper from parasternal short-axis view
  5. 2-d caliper from any other view
LV mass index (LVMI; g/m^2) | 6 months (optional, personalized) and 12 months
  Calculated by the following measurements based on echocardiography.
  Equation: LVMI = LV mass / BSA
  * {(0.8 * [1.04 * ((LVEDD + IVSd + PWd)^3 - LVEDD^3)]) + 0.6} / BSA
  IVSd: Interventricular septum dimension (mm)* PWd: LV Posterior wall dimension (mm)* BSA: body surface area (kg/m^2) calculated from weight (kg) and height (m) at the timing of echocardiography (BSA = weight/ (height)^2
  * LVEDD, IVSd, PWd are measured with the following priority
  1. M-mode from parasternal long-axis view
  2. 2-d caliper from parasternal long-axis view
  3. M-mode from parasternal short-axis view
  4. 2-d caliper from parasternal short-axis view
  5. 2-d caliper from any other view
Left atrial volume index (LAVI, ml/m^2) | 6 months (optional, personalized) and 12 months
  LAVI = LA volume (ml) /BSA (m^2)
  1. LA volume is measured by the biplane area-length method in the apical 4-chamber and apical 2-chamber view as described in:
     (Eur J Echocardiogr. 2008 May;9(3):351-5. doi: 10.1016/j.euje.2007.05.004. Epub 2007 Jul 23.) LA volume = (0.85 × A1 × A2)/(L1 -L2 /2).
  2. BSA: body surface area (kg/m^2) calculated from weight (kg) and height (m) at the timing of echocardiography (BSA = weight/ (height)^2
E/E' ratio | 6 months (optional, personalized) and 12 months
  measurements based on echocardiography E: by pulsed wave Doppler of mitral inflow velocity E': by tissue Doppler of early diastolic mitral annulus velocity
Right ventricular systolic pressure (RVSP, mmHg) | 6 months (optional, personalized) and 12 months
  Right ventricular systolic pressure (RVSP) estimated by Tricuspid valve Regurgitation jet maximum velocity (TR Vmax) base on continuous wave Doppler echocardiographic measurements.
  Modified Bernoulli equation: RVSP = 4V^2 + RA pressure(*)
  * RA pressure (mmHg) is estimated by the following:
  1. RAP=5 when inferior vena cava (IVC) diameter =< 2.1cm and abscent plethora
  2. RAP=10 when IVC =< 2.1cm and present plethora
  3. RAP=10 when IVC > 2.1cm and abscent plethora
  4. RAP=15 when IVC > 2.1cm and present plethora.
LV 4-dimensional strain (percent) | 6 months (optional, personalized) and 12 months
  Using a Vivid E9, E90, E95 ultrasound system (GE Healthcare, Chicago, IL, USA) with a 2.5-3.6 MHz 4-dimensional Volume transducer, a 4D full-volume scan is obtained from the apical position during an end-expiratory apnea. From a twelve-slice display mode, the examiner ensures that the whole LV structure be included in the 4D full-volume image. The frame rate was required to be over 40 percent of the heart rate (HR). The global strain values, including LV GLS, GRS, GCS, and GAS, were automatically calculated by the software. Specific techniques are described in (Eur J Echocardiogr. 2011 Jan;12(1):26-32. doi: 10.1093/ejechocard/jeq095. Epub 2010 Aug 24.)
  * GLS = global longitudinal strain; GRS = global radial strain; GCS = global circumferential strain; GAS = global area strain;
Change in hemoglobin (g/dL) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in albumin (g/dL) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in total bilirubin (mg/dL) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in fasting blood glucose (mg/dL) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in blood urea nitrogen (mg/dL) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in creatinine (mg/dL) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in estimated GFR (ml/min/1.73m^2) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods Calculated by CKD-EPI equation
  CKD-EPI eGFR(mL/min/1.73m^2) = A × (Scr/B)^C × 0.993^(age) , where A, B, and C are the following:
  Female Scr ≤0.7; A = 144, B = 0.7, C = -0.329 Scr ≤0.9; A = 141, B = 0.9, C = -0.411
  Male Scr >0.7; A = 144, B = 0.7, C = -1.209 Scr >0.9; A = 141, B = 0.9, C = -1.209
Change in sodium (mmol/L) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in potassium (mmol/L) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Change in hemoglobin A1c (percent) | Baseline, 6 months and 12 months
  Changes in laboratory values between time periods
Reason for discontinuation of study drug | 6 months and 12 months
  Choose one answer from the following:
  1. cardiogenic shock: persistent hypotension (SBP<90mmHg or MAP drop 30mmHg) with cardiac index < 1.8L/min/m2 without support (< 2.2 with support)
  2. noncardiogenic shock: persistent hypotension and inadequate tissue perfusion(*) excluding cardiac origin
  3. drug intolerance - 'orthostatic hypotension' or 'others'
  4. renal dysfunction (**)
  5. switch to other RAS blocker - specify reason in free text
  6. decision for other advanced cardiac treatment: left ventricular assist device, heart transplantation.
  7. others (free text)
  [*] Shock as defined in (N Engl J Med 2013; 369:1726-1734). [**] Renal dysfunction defined as:
  1. Acute kidney injury (AKI) by KDIGO (Kidney Int Suppl. 2012;2(Suppl 1):8.)
  2. Progression of CKD defined as: sustained reduction in eGFR by 15 mL/min/1.73 m2 (or CKD stage change), or to <10 mL/min/1.73 m2 (or initiation of dialysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The access criteria has not been discussed yet.

REFERENCES:
- [Background] Halliday BP, Wassall R, Lota AS, Khalique Z, Gregson J, Newsome S, Jackson R, Rahneva T, Wage R, Smith G, Venneri L, Tayal U, Auger D, Midwinter W, Whiffin N, Rajani R, Dungu JN, Pantazis A, Cook SA, Ware JS, Baksi AJ, Pennell DJ, Rosen SD, Cowie MR, Cleland JGF, Prasad SK. Withdrawal of pharmacological treatment for heart failure in patients with recovered dilated cardiomyopathy (TRED-HF): an open-label, pilot, randomised trial. Lancet. 2019 Jan 5;393(10166):61-73. doi: 10.1016/S0140-6736(18)32484-X. Epub 2018 Nov 11. PMID 30429050
- [Background] Januzzi JL Jr, Prescott MF, Butler J, Felker GM, Maisel AS, McCague K, Camacho A, Pina IL, Rocha RA, Shah AM, Williamson KM, Solomon SD; PROVE-HF Investigators. Association of Change in N-Terminal Pro-B-Type Natriuretic Peptide Following Initiation of Sacubitril-Valsartan Treatment With Cardiac Structure and Function in Patients With Heart Failure With Reduced Ejection Fraction. JAMA. 2019 Sep 17;322(11):1085-1095. doi: 10.1001/jama.2019.12821. PMID 31475295
- [Background] Wilcox JE, Fang JC, Margulies KB, Mann DL. Heart Failure With Recovered Left Ventricular Ejection Fraction: JACC Scientific Expert Panel. J Am Coll Cardiol. 2020 Aug 11;76(6):719-734. doi: 10.1016/j.jacc.2020.05.075. PMID 32762907
- [Derived] Bak M, Park Y, Kim D, Shin H, Hong D, Yang JH, Choi JO. Angiotensin receptor blocker versus angiotensin receptor-neprilysin inhibitor in improved HF with stabilized NT-proBNP levels. Rev Esp Cardiol (Engl Ed). 2025 Dec 11:S1885-5857(25)00350-0. doi: 10.1016/j.rec.2025.12.006. Online ahead of print. English, Spanish. PMID 41390047